CLINICAL TRIAL: NCT05366764
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of SAR443765 in Healthy Adult Participants and of a Single Dose of SAR443765 in Participants With Mild-to-moderate Asthma
Brief Title: First-in-human Study of SAR443765 in Healthy Participants and in Asthmatic Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDY16622; U1111-1265-6232 (Registry Identifier: ICTRP); PDY16622 (Other: Sanofi Identifier); 2021-000356-19 (EudraCT Number)
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAR443765 (Experimental): Single dose administration of SAR443765
  Interventions: Drug: SAR443765; Drug: Salbutamol or levosalbutamol
- Placebo (Placebo Comparator): Placebo to match SAR443765
  Interventions: Drug: Placebo; Drug: Salbutamol or levosalbutamol

INTERVENTIONS:
Drug: SAR443765 — solution for injection
  Arms: SAR443765
Drug: Placebo — solution for injection
  Arms: Placebo
Drug: Salbutamol or levosalbutamol — metered dose inhaler

SUMMARY:
This is a 3-part, parallel group treatment, Phase 1, randomized, double-blind, placebo-controlled study to assess the safety, tolerability and pharmacokinetics after sequential single and multiple ascending doses of SAR443765 in healthy adult participants, and after a single dose of SAR443765 in participants with mild-to-moderate asthma.

DETAILED DESCRIPTION:
The anticipated study duration per participant is up to 14 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma for at least 12 months and confirmed at screening based on the Global Initiative for Asthma (GINA) 2020 Guidelines
* Controlled asthma defined as no more than 1 canister of rescue inhaler per month over the last 3 months prior to baseline
* Elevated FeNO level defined as ≥25 ppb
* Participants, using as-needed SABA, ICS-naïve or with existing stable treatment (at least for 3 months prior to screening) with low to medium daily dose ICS (≤500 mcg of fluticasone propionate or comparable ICS daily dosage) potentially in combination with a LABA and/or LAMA as second controller, and/or with stable daily leukotriene receptor antagonist, leukotriene synthesis inhibitor and/or chromones
* Prebronchodilator forced expiratory volume in 1 second (FEV1) ≥60% of predicted normal
* Reversibility of at least 12% and 200 mL in FEV1 or forced vital capacity (FVC) after administration of 4 puffs (400 mcg) of albuterol/salbutamol or levalbuterol/levosalbutamol during screening or documented history of a reversibility test that meets this criteria within 5 years prior to screening or documented positive response to methacholine challenge (a decrease in FEV1 by 20% [PC20] of <8 mg/mL) within 5 years prior to screening visit
* Body weight between 50.0 and 105.0 kg, inclusive, if male, and between 40.0 and 95.0 kg, inclusive, if female, body mass index between 18.0 and 32.0 kg/m2
* Male participants are eligible to participate if they use condom during study period
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies: Is a woman of non-childbearing potential (WONCBP) OR Is a woman of childbearing potential (WOCBP) and agrees to use a contraceptive method that is highly effective
* A WOCBP must have a negative highly sensitive pregnancy test within 36 hours before the first administration of study intervention

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any clinically relevant abnormal findings in medical history, physical examination, vital signs, 12-lead ECG.
* Chronic lung disease, or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* History of life-threatening asthma, asthma exacerbation or use of systemic steroid within 3 months prior to screening visit
* Worsening of asthma or respiratory infection within the last 6 weeks prior screening visit.
* Symptomatic postural hypotension,history or presence of drug or alcohol abuse, current smoker or previous smoker with a smoking history >10 pack-years.
* Excessive consumption of beverages containing xanthine bases (more than 4 cups or glasses per day).

NOTE: Other Inclusion/Exclusion criteria may apply. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) /TEAEs | From baseline up to Day 71
  Incidence of adverse events (AEs) and treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Pharmacokinetic (PK) assessment: Cmax | From baseline up to Day 71
  Observed maximum plasma concentration
Pharmacokinetic (PK) assessment: AUClast | From baseline up to Day 71
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time tlast
Pharmacokinetic (PK) assessment: AUC | From baseline up to Day 71
  Area under the serum concentration versus time curve extrapolated to infinity
Change in Nitric Oxide (FeNO) level | Day 1 and Day 29
  Change from Baseline in FeNO level at Day 29
Presence of Anti-SAR443765 antibodies (ADA) | From baseline up to Day 71
  Number of participant with SAR443765 antibodies
Total (free + bound) serum target concentrations of TSLP | From baseline up to Day 71
  Change from baseline in total serum target concentrations of TSLP
Total (free + bound) serum target concentrations of IL-13 | From baseline up to Day 71
  Change from baseline in total serum target concentrations of IL-13

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- Investigational Site Number : 2760001, Berlin, Germany
- Investigational Site Number : 8260001, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Deiteren A, Krupka E, Bontinck L, Imberdis K, Conickx G, Bas S, Patel N, Staudinger HW, Suratt BT. A proof-of-mechanism trial in asthma with lunsekimig, a bispecific NANOBODY molecule. Eur Respir J. 2025 Apr 24;65(4):2401461. doi: 10.1183/13993003.01461-2024. Print 2025 Apr. PMID 39884759
- [Derived] Deiteren A, Bontinck L, Conickx G, Vigan M, Dervaux N, Gassiot M, Bas S, Suratt B, Staudinger H, Krupka E. A first-in-human, single and multiple dose study of lunsekimig, a novel anti-TSLP/anti-IL-13 NANOBODY(R) compound, in healthy volunteers. Clin Transl Sci. 2024 Jun;17(6):e13864. doi: 10.1111/cts.13864. PMID 38924698
- See also: PDY16622 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25316&tenant=MT_SNY_9011